CLINICAL TRIAL: NCT00608972
Title: A Phase II Trial of Doxil, Carboplatin and Bevacizumab in Triple Negative Previously Untreated Metastatic Breast Cancer
Brief Title: Phase II Trial of Doxil, Carboplatin, Bevacizumab in Triple Negative Untreated Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Deborah Toppmeyer, MD, Professor, CINJ, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040702; NJ 2107; Pro0220070274 (Other: CINJ); P30CA072720 (NIH); NCI-2012-00524 (Other: NCI)
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Breast Cancer
Keywords: negative for a protein called HER2/neu; negative for estrogen receptors (ER) and progesterone receptors (PR).; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxil, Carboplatin and Bevacizumab (Experimental)
  Interventions: Drug: Doxil; Drug: Carboplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Doxil — Doxil 30 mg/m2 will be administered on Day 1 of each 28-day cycle.
Drug: Carboplatin — Carboplatin 30 mg/m2 will be administered on Day 1 of each 28-day cycle.
Drug: Bevacizumab — Bevacizumab 10 mg/kg will be administered on Day 1 immediately following chemotherapy and alone on Day 15 of each 28-day cycle.
  Other Names: Avastin

SUMMARY:
The purpose of this research study is to look at the effectiveness of a combination of doxil, carboplatin and bevacizumab on metastatic breast cancer. The type of breast cancer being studied is negative for a protein called HER2/neu and for estrogen receptors (ER) and progesterone receptors (PR). HER2/neu, ER and PR are part of a family of receptors found on both cancer and normal cells. This family of receptors is important for cell growth and is found in many tumor types.This study is being conducted for the following research purposes:· To find out what effects, if any, the study drug has on metastatic breast cancer. For instance, will the study drug cause the tumor(s) to shrink or stop growing?· To test the safety of the study drugs and to see what affects it has. For instance, are there any side effects? If so, what kind of side effects does the study drug cause? How severe are the side effects, and how often do they occur?· To see if the study drugs have any effect on keeping the disease from getting worse.

ELIGIBILITY:
Inclusion Criteria:

1. Women with previously untreated metastatic breast cancer, ER/PR/HER2/neu negative.
2. Age >= 18
3. ECOG performance status <= 2
4. Normal organ and marrow function
5. Normal cardiac function as evidenced by LVEF within institutional normal limits

Exclusion Criteria:

1. History of hypersensitivity reactions to doxil or bevacizumab
2. Myocardial infarct or unstable angina within 6 months before enrollment
3. Prior anthracycline dose exceeding 360 mg/m2 for doxorubicin (including DOXIL) or 720 mg/m2 for epirubicin.
4. Proteinuria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-05-16 (Actual); Primary Completion 2015-07-12 (Actual); Study Completion 2015-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Toppmeyer, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (7):
- United States (7):
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Overlook Medical Center, Summit, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ICH GCP Clinical Trials Registry — https://ichgcp.net/clinical-trials-registry/NCT00608972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Rutgers Cancer Institute of New Jersey Oncology Group. They study was open to accrual on 05/16/2008 and closed to accrual on 12/31/2012.
Pre-assignment Details: We are reporting results on 31 eligible patients.
Period: Overall Study
Arm/Group | Doxil, Carboplatin and Bevacizumab
Started | 31
Completed | 2
Not Completed | 29

BASELINE CHARACTERISTICS:
Arm/Group | Doxil, Carboplatin and Bevacizumab
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) After Treatment With Doxil, Carboplatin and Bevacizumab in Patients With ER, PR, HER2neu Negative Metastatic Breast Cancer
Time Frame: Two Years
Measure: Number; unit: participants
Arm/Group | Doxil, Carboplatin and Bevacizumab
Number analyzed (Participants) | 31
participants | 6

2. Secondary Outcome: Clinical Benefit Rate (CBR=CR+PR+SD)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: up to two years
Measure: Count of Participants; unit: Participants
Arm/Group | Doxil, Carboplatin and Bevacizumab
Number analyzed (Participants) | 31
Participants | 13

3. Secondary Outcome: One-year Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: one year
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Doxil, Carboplatin and Bevacizumab
Number analyzed (Participants) | 31
participants | 31 [29.5 to 65.1]

4. Secondary Outcome: Median Overall Survival After Treatment With Doxil, Carboplatin and Bevacizumab in Patients With ER, PR, HER2neu Negative
Description: median overall survival
Time Frame: From date of randomization up to two years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Doxil, Carboplatin and Bevacizumab
Number analyzed (Participants) | 31
months | 11 [8.8 to 21.8]

5. Secondary Outcome: Six-month Survival After Treatment With Doxil, Carboplatin and Bevacizumab in Patients With ER, PR, HER2neu Negative
Description: Six-month survival rate
Time Frame: six months
Measure: Number (95% Confidence Interval); unit: Percentage participants
Arm/Group | Doxil, Carboplatin and Bevacizumab
Number analyzed (Participants) | 31
Percentage participants | 41.9 [24.6 to 59.3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 913 days per patient.
Arm/Group | Doxil, Carboplatin and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 28/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol: Protocol #1 (2013-10-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT00608972/Prot_000.pdf
  • Study Protocol: Protocol #2 (2013-10-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT00608972/Prot_001.pdf
  • Study Protocol and Statistical Analysis Plan: Protocol #4SAP (2013-10-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT00608972/Prot_SAP_002.pdf
  • Informed Consent Form (2011-10-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT00608972/ICF_003.pdf